CLINICAL TRIAL: NCT04003779
Title: Reconfiguring the Patient Room for a Fall Protection Strategy to Increase Patient Stability During Ambulation
Brief Title: Reconfiguring the Patient Room to Increase Patient Stability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: The Center for Health Design (Unknown)
Responsible Party: Principal Investigator, Bob Wong, Professor, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 00099410
Record Dates: First submitted 2019-06-25; First posted 2019-07-01 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Elderly, Frail; Accidental Falls; Hospitals

STUDY DESIGN:
Intervention Model Description: Using virtual reality and ergonomic measures, we will sequentially adjust features of the hospital room to determine the most stable gate in frail elderly patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participant stability with various room configurations (Other): Single-arm. Ergonomically exploring patient stability moving around various configurations of a hospital room.
  Interventions: Other: Room configuration

INTERVENTIONS:
Other: Room configuration — Adjust distance, handrails, degrees of turn for participant

SUMMARY:
Despite decades of research into patient falls, falls and the injuries incurred continue to be a serious threat to patient safety. Fall rates continue to be unacceptably high. The purpose of this project is to increase the safety of a hospital room for patient mobility, using innovative simulation strategies and patient-centric design.

DETAILED DESCRIPTION:
Despite decades of research into patient falls, falls and the injuries incurred continue to be a serious threat to patient safety. Fall rates continue to be unacceptably high. The purpose of this project is to increase the safety of a hospital room for patient mobility, using innovative simulation strategies and patient-centric design.

An innovative simulation environment will be built to enable rapid assessment of room layout and fixture positioning and patient stability. The results from multiple simulations will be used to fabricate a prototype room layout that will be tested by patients with Parkinson disease and reviewed and updated with input from other relevant stakeholders. A final room prototype will be built and tested. Results will be translated and shared with all stakeholders and disseminated for implementation.

ELIGIBILITY:
Inclusion Criteria:

* Frail elderly, impaired gait

Exclusion Criteria:

* Use of walking aid

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-07-14 (Actual); Primary Completion 2024-09-29 (Actual); Study Completion 2024-09-29 (Actual)

PRIMARY OUTCOMES:
Gait: increased stability | 24 months
  Increased balance

CONTACTS AND LOCATIONS:
Overall Officials: Bob G Wong, PhD, Principal Investigator — University of Utah; Andrew Merryweather, PhD, Principal Investigator — University of Utah
Locations (1):
- Dumke Health Professions Building, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No